CLINICAL TRIAL: NCT05678595
Title: The Effect of High-intensity Laser Therapy on Pain, Functional Status, Hand Grip Strength and Median Nerve Cross-sectional Area in Ultrasonography in Patients With Carpal Tunnel Syndrome.
Brief Title: The Effect of High-intensity Laser Therapy in Patients With Carpal Tunnel Syndrome.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Banu Ordahan, Clinical Professor, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: fatih yiğit
Record Dates: First submitted 2023-01-02; First posted 2023-01-10 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Carpal Tunnel Syndrome
Keywords: pain; High-intensity laser therapy; ultrasonography
MeSH Terms: conditions — Carpal Tunnel Syndrome; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A hot laser derived from a Nd: YAG laser (Active Comparator): HILT: A hot laser derived from a Nd: YAG laser has 12 W (watt) and 1064 nm characteristics. The device will administered to the hand wrist area in two steps in the HILT group: phase I and phase II. The application will made utilizing continuous circular movements in both phases I and II. The first five sessions consisted of a 100-second intermittent phase analgesic effect at 8 W and 8 J/cm2 for a total energy of 200 J. The following five sessions consisted of a continuous 11 minutes 6 second bio stimulating effect with a dosage of 3 W 80 J/cm2. Over the course of two weeks, ten treatment sessions of HILT will be given.
  Interventions: Device: high-intensity laser therapy; Device: sham high-intensity laser therapy
- sham high-intensity laser therapy (Sham Comparator): HILT is administered as a placebo for two weeks, 5 sessions a week, for a total of 10 sessions.
  Interventions: Device: high-intensity laser therapy; Device: sham high-intensity laser therapy

INTERVENTIONS:
Device: high-intensity laser therapy — HILT: A hot laser derived from a Nd: YAG laser has 12 W (watt) and 1064 nm characteristics. The device will administered to the hand wrist area in two steps in the HILT group: phase I and phase II. The application will made utilizing continuous circular movements in both phases I and II. The first five sessions consisted of a 100-second intermittent phase analgesic effect at 8 W and 8 J/cm2 for a total energy of 200 J. The following five sessions consisted of a continuous 11 minutes 6 second bio stimulating effect with a dosage of 3 W 80 J/cm2. Over the course of two weeks, ten treatment sessions of HILT will be given.
Device: sham high-intensity laser therapy — HILT is administered as a placebo for two weeks, 5 sessions a week, for a total of 10 sessions.

SUMMARY:
The aim of this study is to evaluate the effects of high intensity laser therapy (HILT) on pain, functional status, hand grip strength and median nerve cross-sectional area in ultrasonography in patients with carpal tunnel syndrome.

DETAILED DESCRIPTION:
Patients who are admitted and diagnosed with carpal tunnel syndrome based on anamnesis, physical examination and electromyography are included in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Electrophysiologically mild or moderate CTS
2. Patients who are literate and able to understand verbal instructions in our

Exclusion Criteria:

1. Diabetes
2. Systemic disorders that may affect treatment such as hypothyroidism, SLE, gout
3. History of polyneuropathy, cervical radiculopathy, brachial plexopathy
4. Injection for the carpal tunnel in the last 1 month
5. History of severe trauma, fracture, operation to both upper extremities at any time
6. Malignancy or history of malignancy
7. Renal failure
8. Peripheral or central nervous system diseases
9. Pregnancy
10. History of physical therapy program for the same hand wrist in the last months.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-06-23 (Actual); Study Completion 2023-06-23 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | Change from baseline in pain on the VAS at week 2 and week 12 [ Time Frame: Baseline-Week 2- Week 12 ]
  Visual Analog Scale (VAS) is used to measure and monitor the intensity of pain.

SECONDARY OUTCOMES:
Boston Carpal Tunnel Questionnaire | Change from baseline in pain and disability on the Boston Carpal Tunnel Questionnaire at week 2 and 12.
  The Boston Carpal Tunnel Score is a patient-reported questionnaire that examines symptom severity and overall functional status of patients with carpal tunnel syndrome. The Symptom Severity Scale (SSS) with 11 questions is scored on a Likert scale of 1-5 and the Functional Status Scale (FSS) with 8 questions is scored from 1-5 with 1 as no difficulty and 5 as difficult.
Hand Grip Force Measurement Test | Baseline- week 2- week 12
  A hydraulic hand dynamometer (Jamar) will be used in the measurements. Three measurements will be made with the elbow flexed and connected to the body, and the forearm in a neutral position. The measurements will be averaged in kg-f and recorded in the study form.
The cross-sectional area of the median nerve | Change from baseline in the cross-sectional area of the median nerve at week 2 and week 12.
  The cross-sectional area of the median nerve will be measured by USG at the level of the pisiform bone (proximal carpal tunnel). While the patient is in a sitting position, the arm on the measuring side will be positioned semiflexed, elbow semiflexed, forearm supinated, fingers semi-flexed, and wrist on a flat surface.

CONTACTS AND LOCATIONS:
Overall Officials: BANU ORDAHAN, Principal Investigator — Meram Medical School, Necmettin Erbakan University, Konya, Turkey
Locations (1):
- Banu Ordahan, Konya, Turkey (Türkiye)